CLINICAL TRIAL: NCT06379321
Title: A Retrospective/Prospective, Post-market, Multi-center Evaluation of the Clinical Outcomes of the Triathlon Hinge Knee (THK) System
Brief Title: Evaluation of Outcomes of the Triathlon Hinge Knee (THK) System
Acronym: Hinge
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-362
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Knee Arthropathy; Recurrence; Knee Infection
MeSH Terms: conditions — Recurrence | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Primary: Triathlon Hinge Femoral Component + Revision Baseplate
  Interventions: Device: Triathlon Hinge Knee (THK) System
- Revision: Triathlon Hinge Femoral Component+ Revision Baseplate
  Interventions: Device: Triathlon Hinge Knee (THK) System
- TS Revision: Triathlon TS Femoral Component+ Revision Baseplate
  Interventions: Device: Triathlon Hinge Knee (THK) System
- Revision (Maximum of 80 subjects): Triathlon TS Femoral Component + Revision Baseplate
  Interventions: Device: Triathlon Hinge Knee (THK) System
- MRH Revision: MRH Femoral Component + Revision Baseplate
  Interventions: Device: Triathlon Hinge Knee (THK) System
- GMRS Primary or Revision: GMRS Femoral Component + Revision Baseplate
  Interventions: Device: Triathlon Hinge Knee (THK) System

INTERVENTIONS:
Device: Triathlon Hinge Knee (THK) System — Participants receive Triathlon Hinge Knee (THK) System during primary or revision knee arthroplasty in accordance with the indications for use

SUMMARY:
This study is a prospectively and retrospectively enrolled, post-market, open-label, non-randomized, single institution evaluation of clinical outcomes of primary or revision knee surgery patients who meet the eligibility criteria and received devices from the Triathlon Hinge Knee System according to its indications for use (IFU).

Clinical evaluation for all cases will include data collection of patient demographics, surgical details, early postoperative status, functional and clinical outcomes, and survivorship at 1, 2, 6, and 10-years.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and performance of the Triathlon Hinge Knee System for both primary and revision cases in accordance with the Indications for Use.

The main objective of this study is to determine (1) mid- (5 year) and long-term (10 year) survivorship, and (2) drivers of failure for the THK hinge. Data from this study will be used to develop a predictive model to identify the most important factors in achieving fixation, including the role of augments, cones, thresholds for cement mantle thickness, and number of zones of fixation required for survivorship.

Survivorship is defined as the absence of aseptic revision to the implanted device.

The Triathlon Hinge Knee System consists of Triathlon Hinge femoral components, the Triathlon Revision baseplate, Triathlon Revision Tibial Augments, Triathlon Hinge Femoral Distal Augments, Triathlon Hinge Insert, Triathlon Revision Insert X3, and Triathlon Hinge Bumpers, Axle, Bushings, Tibial Sleeve, and Bearing component.

It is designed to be a single platform for revision, difficult primary, and limb salvage surgeries.

ELIGIBILITY:
Inclusion Criteria:

* The subject undergoes a primary or revision procedure implanting at least the Revision Baseplate portion of the Triathlon Hinge Knee System in accordance with the Indications for Use.
* The subject has signed an IRB/EC-approved, study-specific Informed Consent Form (ICF).
* The subject is a male or non-pregnant female at the time of enrollment.
* The subject agrees to comply with the protocol-mandated clinical evaluations.

Exclusion Criteria:

* Any active or suspected latent infection in or about the knee joint; overt infection;
* Distant foci of infection which may cause hematogenous spread to the implant site; rapid disease progression as manifested by joint destruction or bone resorption apparent on roentgenogram;
* skeletally immature patients;
* Severe instability of the knee joint secondary to the absence of collateral ligament integrity and function.
* Bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* Known or suspected sensitivity and/or allergy to any material in the device.
* Conditions presenting an increased risk of failure include:
* uncooperative patient or patient with neurologic disorder, incapable of following instructions;
* osteoporosis;
* metabolic disorders which may impair bone formation or cause bone loss;
* osteomalacia; and,
* previous arthrodesis.
* A higher incidence of implant failure has also occurred in paraplegics, cerebral palsy and patients with Parkinson's disease.
* Any mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The subject is a prisoner

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants who meet the eligibility criteria and receive/received devices from the Triathlon Hinge Knee System according to its indications for use (IFU).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2034-05-10 (Estimated); Study Completion 2034-05-10 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 1, 2, 6 and 10 years
  To evaluate the survivorship of the Hinge Knee System at postoperatively. Survival is defined as the absence of aseptic revision to the implanted device.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Deren, M.D., Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No